CLINICAL TRIAL: NCT03920098
Title: The Chilean Maternal and Infant Nutrition Cohort Study II
Brief Title: Chilean Maternal & Infant Cohort Study II (CHiMINCs-II)
Acronym: CHiMINCs-II
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Instituto de Nutrición y Tecnología de los Alimentos (Other)
Collaborators: Pontificia Universidad Catolica de Chile (Other); Servicio de Salud Metropolitano Sur Oriente (Other Government)
Responsible Party: Principal Investigator, Dr. Maria Luisa Garmendia, Associate Professor, Instituto de Nutrición y Tecnología de los Alimentos
Other Study IDs: 1190532
Record Dates: First submitted 2019-04-16; First posted 2019-04-18 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Breast Density; Body Composition; Nutritional Status; Mental Health Issue
Keywords: Breast densities; Breast neoplasms; Glucose metabolism disorders; Diabetes, gestational; Pregnancy; Nutritional status; Mental health; Body composition; Growth and development; Primary Health Care; Dual-energy X-ray Absorptiometry; Latin America; Chile
MeSH Terms: conditions — Breast Neoplasms; Glucose Metabolism Disorders; Diabetes, Gestational; Psychological Well-Being | interventions — Nutritional Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Additional fasting venous samples will be collected during routine public health care blood extractions and at delivery (maternal venous and umbilical cord blood samples). Also, feces samples of newborn will be collected after delivery. Whole blood, plasma, buffy coat, serum and red blood cells will be separated by centrifugation within the next 3 hours. Biological specimens will be aliquot and keep to -80ºC until the determination of metabolic markers, growth factors and hormones.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mother-infant dyads: Mother-infant dyads
  Interventions: Other: Nutrition and mental health during pregnancy

INTERVENTIONS:
Other: Nutrition and mental health during pregnancy — Altered metabolic milieu is defined as a fasting glucose level >100 mg/dL at the first trimester of pregnancy by national guidelines. Altered metabolic milieu during the second trimester (24-28 weeks of pregnancy) is defined as a fasting glucose levels > 92 mg/dL and/or plasma glucose levels > 153 mg/dL two hours after load in the oral glucose tolerance test according to ADA guidelines or a fasting glucose >100 mg/dL and/or > 140 mg/dL two hours after load in the oral glucose tolerance test according to national guidelines. The COVID-19 pandemic is considered as a natural nutritional and mental health exposure.

SUMMARY:
The Chilean Maternal & Infant Cohort Study II (ChiMINCs II) is an ongoing cohort that is part of the Chilean Maternal and Infant Nutrition Observatory of the South-East area of Santiago, Chile. In total, 1927 pregnant women beneficiaries of the public health systems and their offspring were recruited before 12 weeks of gestation and are followed across pregnancy (<15, 26-28, and 35-37 weeks of gestation) and up to 2 years of age of their offspring. Two studies are currently nested in ChiMINCs II: 1) Breast Cancer Risk Assessment in Mothers (BRECAM) study, and 2) the ChiMINCs-COVID study. The primary objective of BRECAM study is to test the association between maternal metabolic indicators (i.e., insulin, glucose, IGF-1, and HbAc1 concentrations) at early pregnancy (i.e., <15 and 26-28 weeks of gestation) and breast density 3 months after the cessation of lactation. For this purpose, we collect maternal obstetric, lifestyle, dietary intake, anthropometric, and biochemical information. The aim of the ChiMINCs-COVID study is to assess dietary-related risks and mental health problems derived from the COVID-19 pandemic and their influence on maternal and infant's health and nutrition. Thus, we collected detailed information on dietary behaviors, mental health and COVID-related information at each trimester, along with neonatal and infant nutritional information. The purpose of the present work is to describe the design, methods, and descriptive information at recruitment of ChiMINCs-II, also discussing the implications that this study can have to better understand maternal and infant nutrition and health during the COVID-19 era.

ELIGIBILITY:
Inclusion Criteria:

* 18 or more years of age
* Gestation <15 weeks at first prenatal visit
* No intention to move outside the city of Santiago in the next to years

Exclusion Criteria:

* High-risk pregnancy (i.e., preeclampsia, pre- existing diabetes)
* Pre-existing cancer or family history of breast cancer
* Intended to migrate from the public to the private health care system

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Study Population: We identified pregnant women who received primary prenatal care within PHCC located in the South East area of Santiago. After, offspring of pregnant women were followed postnatally.
Sampling Method: Probability Sample
Enrollment: 1927 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-07-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Breast absolute (AFGV) fibro-glandular volume measured by DXA technique | Three months after breastfeeding cessation
  cm3
Breast absolute percentage (%FVG) of fibro-glandular volume measured by DXA technique | Three months after breastfeeding cessation
  percentage
Gestational weight gain | At delivery
  kg
Gestational Diabetes | At delivery
  Percentage of mothers diagnosed
Pregnancy Risk Assessment Monitoring System | Through the gestation, up the delivery
  Score
Edinburg Postnatal Depression Scale | Through the gestation, up to 6 months
  Score
Glucose concentration | Through the gestation, up the delivery
  mg/dL
Insulin concentration | Through the gestation, up the delivery
  uIU/mL
Pandemic Anxiety Scale | Through the gestation, up the delivery
  Score

SECONDARY OUTCOMES:
Offspring weight | At 6 months of age
  g
Offspring length | At 6 months of age
  cm
Offspring head circumference | At 6 months of age
  cm
Offspring body fat | At 6 months of age
  Percentage

CONTACTS AND LOCATIONS:
Overall Officials: María L Garmendia, PhD, Principal Investigator — Instituto de Nutrición y Tecnología de Alimentos; Camila L Corvalán Aguilar, PhD, Principal Investigator — Institute of Nutrition and Food Technology (INTA), University of Chile, Chile; María F Mujica Coopman, PhD, Principal Investigator — Institute of Nutrition and Food Technology (INTA), University of Chile, Chile
Locations (1):
- Corporación de Salud Municipal de Puente Alto, Santiago, Puente Alto, Chile

IPD SHARING:
Plan to Share IPD: No
Data and blood samples that will be collected in this study will be under the custody of the principal investigator and a human subject protection review board will regulate its use. Others researchers may access the data by contacting to María Luisa Garmendia (Principal Investigator).

REFERENCES:
- [Background] McCormack VA, dos Santos Silva I. Breast density and parenchymal patterns as markers of breast cancer risk: a meta-analysis. Cancer Epidemiol Biomarkers Prev. 2006 Jun;15(6):1159-69. doi: 10.1158/1055-9965.EPI-06-0034. PMID 16775176
- [Background] Boyd NF, Guo H, Martin LJ, Sun L, Stone J, Fishell E, Jong RA, Hislop G, Chiarelli A, Minkin S, Yaffe MJ. Mammographic density and the risk and detection of breast cancer. N Engl J Med. 2007 Jan 18;356(3):227-36. doi: 10.1056/NEJMoa062790. PMID 17229950
- [Background] Boyd N, Berman H, Zhu J, Martin LJ, Yaffe MJ, Chavez S, Stanisz G, Hislop G, Chiarelli AM, Minkin S, Paterson AD. The origins of breast cancer associated with mammographic density: a testable biological hypothesis. Breast Cancer Res. 2018 Mar 7;20(1):17. doi: 10.1186/s13058-018-0941-y. PMID 29514672
- [Background] Li T, Sun L, Miller N, Nicklee T, Woo J, Hulse-Smith L, Tsao MS, Khokha R, Martin L, Boyd N. The association of measured breast tissue characteristics with mammographic density and other risk factors for breast cancer. Cancer Epidemiol Biomarkers Prev. 2005 Feb;14(2):343-9. doi: 10.1158/1055-9965.EPI-04-0490. PMID 15734956
- [Background] Boyd NF, Dite GS, Stone J, Gunasekara A, English DR, McCredie MR, Giles GG, Tritchler D, Chiarelli A, Yaffe MJ, Hopper JL. Heritability of mammographic density, a risk factor for breast cancer. N Engl J Med. 2002 Sep 19;347(12):886-94. doi: 10.1056/NEJMoa013390. PMID 12239257
- [Background] Varghese JS, Thompson DJ, Michailidou K, Lindstrom S, Turnbull C, Brown J, Leyland J, Warren RM, Luben RN, Loos RJ, Wareham NJ, Rommens J, Paterson AD, Martin LJ, Vachon CM, Scott CG, Atkinson EJ, Couch FJ, Apicella C, Southey MC, Stone J, Li J, Eriksson L, Czene K, Boyd NF, Hall P, Hopper JL, Tamimi RM; MODE Consortium; Rahman N, Easton DF. Mammographic breast density and breast cancer: evidence of a shared genetic basis. Cancer Res. 2012 Mar 15;72(6):1478-84. doi: 10.1158/0008-5472.CAN-11-3295. Epub 2012 Jan 19. PMID 22266113
- [Background] Nazari SS, Mukherjee P. An overview of mammographic density and its association with breast cancer. Breast Cancer. 2018 May;25(3):259-267. doi: 10.1007/s12282-018-0857-5. Epub 2018 Apr 12. PMID 29651637
- [Background] Rice MS, Rosner BA, Tamimi RM. Percent mammographic density prediction: development of a model in the nurses' health studies. Cancer Causes Control. 2017 Jul;28(7):677-684. doi: 10.1007/s10552-017-0898-7. Epub 2017 May 6. PMID 28478536
- [Background] Yaghjyan L, Colditz GA, Rosner B, Bertrand KA, Tamimi RM. Reproductive factors related to childbearing and mammographic breast density. Breast Cancer Res Treat. 2016 Jul;158(2):351-9. doi: 10.1007/s10549-016-3884-y. Epub 2016 Jun 28. PMID 27351801
- [Background] Rice MS, Bertrand KA, Lajous M, Tamimi RM, Torres G, Lopez-Ridaura R, Romieu I. Reproductive and lifestyle risk factors and mammographic density in Mexican women. Ann Epidemiol. 2015 Nov;25(11):868-73. doi: 10.1016/j.annepidem.2015.08.006. Epub 2015 Aug 29. PMID 26475982
- [Background] Collaborative Group on Hormonal Factors in Breast Cancer. Breast cancer and breastfeeding: collaborative reanalysis of individual data from 47 epidemiological studies in 30 countries, including 50302 women with breast cancer and 96973 women without the disease. Lancet. 2002 Jul 20;360(9328):187-95. doi: 10.1016/S0140-6736(02)09454-0. PMID 12133652
- [Background] Gabrielson M, Chiesa F, Behmer C, Ronnow K, Czene K, Hall P. Association of reproductive history with breast tissue characteristics and receptor status in the normal breast. Breast Cancer Res Treat. 2018 Aug;170(3):487-497. doi: 10.1007/s10549-018-4768-0. Epub 2018 Mar 30. PMID 29603032
- [Background] Britt K, Ashworth A, Smalley M. Pregnancy and the risk of breast cancer. Endocr Relat Cancer. 2007 Dec;14(4):907-33. doi: 10.1677/ERC-07-0137. PMID 18045947
- [Background] Vashi R, Hooley R, Butler R, Geisel J, Philpotts L. Breast imaging of the pregnant and lactating patient: imaging modalities and pregnancy-associated breast cancer. AJR Am J Roentgenol. 2013 Feb;200(2):321-8. doi: 10.2214/ajr.12.9814. PMID 23345353
- [Background] Sabate JM, Clotet M, Torrubia S, Gomez A, Guerrero R, de las Heras P, Lerma E. Radiologic evaluation of breast disorders related to pregnancy and lactation. Radiographics. 2007 Oct;27 Suppl 1:S101-24. doi: 10.1148/rg.27si075505. PMID 18180221
- [Background] Loehberg CR, Heusinger K, Jud SM, Haeberle L, Hein A, Rauh C, Bani MR, Lux MP, Schrauder MG, Bayer CM, Helbig C, Grolik R, Adamietz B, Schulz-Wendtland R, Beckmann MW, Fasching PA. Assessment of mammographic density before and after first full-term pregnancy. Eur J Cancer Prev. 2010 Nov;19(6):405-12. doi: 10.1097/CEJ.0b013e32833ca1f4. PMID 20700056
- [Background] Strange KS, Wilkinson D, Edin G, Emerman JT. Mitogenic properties of insulin-like growth factors I and II, insulin-like growth factor binding protein-3 and epidermal growth factor on human breast stromal cells in primary culture. Breast Cancer Res Treat. 2004 Mar;84(2):77-84. doi: 10.1023/B:BREA.0000018384.64326.dd. PMID 14999138
- [Background] Rosato V, Bosetti C, Talamini R, Levi F, Montella M, Giacosa A, Negri E, La Vecchia C. Metabolic syndrome and the risk of breast cancer in postmenopausal women. Ann Oncol. 2011 Dec;22(12):2687-2692. doi: 10.1093/annonc/mdr025. Epub 2011 Mar 17. PMID 21415236
- [Background] Agnoli C, Berrino F, Abagnato CA, Muti P, Panico S, Crosignani P, Krogh V. Metabolic syndrome and postmenopausal breast cancer in the ORDET cohort: a nested case-control study. Nutr Metab Cardiovasc Dis. 2010 Jan;20(1):41-8. doi: 10.1016/j.numecd.2009.02.006. Epub 2009 Apr 10. PMID 19361966
- [Background] Buschard K, Thomassen K, Lynge E, Vejborg I, Tjonneland A, von Euler-Chelpin M, Andersen ZJ. Diabetes, diabetes treatment, and mammographic density in Danish Diet, Cancer, and Health cohort. Cancer Causes Control. 2017 Jan;28(1):13-21. doi: 10.1007/s10552-016-0829-z. Epub 2016 Nov 10. PMID 27832382
- [Background] Pereira A, Garmendia ML, Uauy R, Neira P, Lopez-Arana S, Malkov S, Shepherd J. Determinants of volumetric breast density in Chilean premenopausal women. Breast Cancer Res Treat. 2017 Apr;162(2):343-352. doi: 10.1007/s10549-017-4126-7. Epub 2017 Jan 28. PMID 28132392
- [Background] Chen YH, Ferguson KK, Meeker JD, McElrath TF, Mukherjee B. Statistical methods for modeling repeated measures of maternal environmental exposure biomarkers during pregnancy in association with preterm birth. Environ Health. 2015 Jan 26;14:9. doi: 10.1186/1476-069X-14-9. PMID 25619201
- [Derived] Mujica-Coopman MF, Corvalan C, Flores M, Garmendia ML. The Chilean Maternal-Infant Cohort Study-II in the COVID-19 Era: A Study Protocol. Front Public Health. 2022 Jul 14;10:904668. doi: 10.3389/fpubh.2022.904668. eCollection 2022. PMID 35910889